CLINICAL TRIAL: NCT04991363
Title: Effect of Using Image Standardization Device for Dental Photography Standerdizatuon in Comparison to Individualized Photography In Vivo Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Ashraf Abou-Bakr, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: oper 123
Record Dates: First submitted 2021-07-14; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Digital Photography; Standardization; ISD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Procedure: Bleaching

INTERVENTIONS:
Procedure: Bleaching — Digital images for each patient will be taken once with the camera fixed on the classic tripod and again when the camera was fixed on the ISD , then horizontal and vertical measurements of the canines will be recorded by using a computer software on the digital images, then bleaching will be fine for all patients, then a second set of images will be taken again with the tripod and then with ISD, then measurements will be repeated and compared with the first set of images
  Other Names: Image standardization; Tripod; ISD

SUMMARY:
This randomized clinical trial aimed to evaluate the effect of Image Standardization Device (ISD) on standardization of clinical images from the same entry point (patient right 45o).

Digital photography is highly important on multiple levels and has become associated with modern dentistry. Its application in dental practice is simple, quick, and extremely useful for procedures documentation, patient education, and conducting clinical research, resulting in several benefits for dentists in the terms of examination, diagnosis, treatment planning, progress and monitoring treatment outcomes. On the other hand, digital photography becomes significant tool for patient reassurance as showing before and after photos of several procedures helps in patient relaxation and understanding from the start, as well as improves the patient-dentist trust.

In the terms of producing decent digital dental photographs, standardization in several aspects of the photographic equipment, environment, and patient position become a critical issue for successful reproducible photographs.

Different standardization methods have been mentioned in the literature, some of them discussed the standardization characteristics in the terms of camera settings and adjustment using tripod only with standardized camera/patient distance, lighting, and background color. Other studies discussed standardization from a different point of view regarding the standardized patient head position and fixed camera/ patient distance using various devices slightly resembles the ISD used in this study.

The methodology of the current study included a total of twenty patients, photographed with ISD taking duplicate photographs and using individualized photography as a control group via conventional Tripod from the same photography point at 45º from the patient's right side to study the effect of the image standardization device in photograph standardization over conventional imaging methods. The Intervention used in this study was bleaching that was done before taking the same photographs once again from the same projections to reproduce the same images using both methods.

The assessment was done by measuring in millimeters the horizontal and vertical measurements of the canine in each patient by using a ruler tool on digital software and comparing them with the reference standard which was the canine's real measurements.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with full set of anterior teeth willing to participate in the study in return to perform dental bleaching procedures

Exclusion Criteria:

* Patients with missing anterior teeth
* Patients with fillings in labial surface of anterior teeth
* Patients with prosthodontics in anterior teeth
* Patients with dental sensitivity
* Patients under 16 years old (bleaching age restrictions)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Standardized digital imaging | 1 month
  Measuring tool is digital softwares to measure the length of the canine before and after bleaching process, from the images captured by the camera was fixed on the classic tripod or the images taken when the camera was fixed on the ISD , canine real measurements are the gold standard , the measuring unit is in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided